CLINICAL TRIAL: NCT04303338
Title: Effectiveness of Adding Neural Tension to Masotherapy in Patients With Parkinson's Disease
Brief Title: Masotherapy With Neural Tension in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/45
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Essential tremor; Neuromuscular Therapy; Massage; Manual Therapy; Neurodynamic
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masotherapy with neural tension (Experimental): The investigators are going to massage the patient´s upper limb applying a radial nerve neural tension. In order to the upper limb should be positioned lowering the scapula, elbow extended, internal rotation glenohumeral, forearm pronation, bend and cubital deviation of the wrist, fingers bended and thumb adduction, and finally glenohumeral abduction.
  Interventions: Procedure: Masotherapy with neural tension and masotherapy with non-neural tension
- Masotherapy with non-neural tension (Active Comparator): The investigators are going to practice a conventional upper limb massage
  Interventions: Procedure: Masotherapy with neural tension and masotherapy with non-neural tension

INTERVENTIONS:
Procedure: Masotherapy with neural tension and masotherapy with non-neural tension — To compare the effectiveness of masotherapy with neural tension and masotherapy with non-neural tension
  Other Names: Neurodynamic

SUMMARY:
The objective of this study is to assess if the masotherapy with neural tension is more effective than non-neural tension to improve and reduce tremor in patients with Parkinson's disease. The project will be carried out in clinics, where both data collection, assessments and scales will be carried out, as well as the plan and intervention in which the neural tension massage therapy of the radial nerve will be applied to the first intervention group; and massage therapy without neural tension in the second group.

DETAILED DESCRIPTION:
In this study the investigators are going to compare the effectiveness of two treatments (masotherapy with neural tension and masotherapy with non-neural tension) in patients with Parkinson disease based on the improved of pain, tremor, functional and life quality.

The investigators are going to divide the number of volunteers in two groups. The first group is going to be treated during 8 weeks with conventional (non-neural tension) masotherapy in the upper limb, the other group is going to be treated with radial neural tension masotherapy during 8 weeks also. To apply the neural tension, the investigators position the patient's upper limb lowering the scapula, elbow extended, internal rotation glenohumeral, forearm pronation, bend and cubital deviation of the wrist, fingers bended and thumb adduction, and finally glenohumeral abduction.

To compare the results between the different groups, the investigators are going to value the patients 4 times, the first one before the beginning of the treatment, the second one and the end of the treatment, the third one after one month completing the treatment, and the last one after three months completing the treatment.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with Parkinson disease in mild or moderate degree.
* Age between 50-80 years old.
* People who can answer the questionnaires without held.
* People who commit to attend the treatment assigned in the study.
* People with tremor that limit his/her functionality or cause discomfort.
* People who is not treated the upper limb

Exclusion Criteria:

* People with mental disease.
* People who do not sign the informed consent.
* People who present comorbidities that can affect the final result of the study.
* People whose medication is modified through the study.
* People who take medication whose secundary effect is the tremor appearance.
* People who is participating in other research studies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Changes in the tremor | Baseline and 1 month after intervention
  Using the Unified Parkinson's Disease Ratin Scale (UPDRS). Each item is scored 0-4 (0= normal; 10= severe affectation) yielding a total between 0 and 159.

SECONDARY OUTCOMES:
Changes in the health-related quality of life: Parkinson Disease Quality of Questionnaire (PDQ-39) | Baseline 8 weeks and 1 month after intervention
  Using the Parkinson Disease Quality of Questionnaire (PDQ-39). Each item is scored 0-4 (0= better life quality; 4= bad life quality) yielding a total between 0 and 156.
Changes in the strength | Baseline 8 weeks and 1 month after intervention
  Using the MicroFet 2 Hoggan
Changes in the manual dexterity | Baseline 8 weeks and 1 month after intervention
  Using the Coin Rotation Task (CRT)
Changes in the pain: Visual Analog Scale (VAS) | Baseline 8 weeks and 1 month after intervention
  Using the Visual Analog Scale (VAS). Each item is scored 0-10 (0= no pain; 10= the major pain that the patient can imagine) yielding a total between 0 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, PhD, Study Director — University of Jaen
Locations (1):
- Physiotherapy clinic, Madrid, Spain